CLINICAL TRIAL: NCT06246266
Title: Effectiveness of Helfer Skin Tap Technique and ShotBlocker Technique in Reducing Pain in Babies Receiving Intramuscular Vaccination
Brief Title: Effectiveness of Helfer Skin Tap Technique and ShotBlocker Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra TURAL BUYUK, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Helfer Skin Tap
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Pain
Keywords: infant; ıntramuscular; vaccine; Helfer Skin Tap Technique; ShotBlocker; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Helfer Skin Tap Technique group (Experimental): Mechanical stimulation given with the Helfer Skin Tap technique during intramuscular vaccine administration will distract the baby's attention.
  Interventions: Procedure: Helfer Skin Tap Technique group
- ShotBlocker Technique group (Experimental): During intramuscular vaccine administration to babies, the injection ShotBlocker Technique will be applied using the ShotBlocker tool (a tool with a "U" appearance, with blunt but not pointed protrusions).
  Interventions: Procedure: ShotBlocker Technique group

INTERVENTIONS:
Procedure: Helfer Skin Tap Technique group — During intramuscular vaccine administration, the muscle will be tapped with the palmar surface of the fingers of the other hand that is not used, with light rhythmic movements, counting for 1-15 seconds. Then, when the muscle is entered with the injection, it will continue to be hit with light rhythmic movements for 1-3 seconds. Thus, the muscle will relax and the fibers around the muscle will be stimulated. Mechanical stimulation given with the Helfer Skin Tap technique during intramuscular vaccine administration will distract the baby's attention.
  Arms: Helfer Skin Tap Technique group
Procedure: ShotBlocker Technique group — The protruding but not sharp surface on the ShotBlocker tool will be placed on the baby's skin before intramuscular vaccine administration.
  Injection will be applied to the middle part of this vehicle, which has a 'U' appearance. This tool, which does not cause any harm to the skin surface, will provide stimulation to the muscle fibers according to the Gate Control Theory related to pain.
  Arms: ShotBlocker Technique group

SUMMARY:
The purpose of this study is to examine the effectiveness of the Helfer Skin Tap Technique and the ShotBlocker Technique in reducing pain in babies receiving intramuscular vaccination.

DETAILED DESCRIPTION:
During immunization, babies feel pain from the injection and give behavioral reactions such as crying and struggling in response to this pain. Pain-reducing methods (Buzzy device, cold application, hot application, music, virtual reality, distracting cards, stress ball, etc.) are used during intramuscular vaccine injection in children. Studies using the Helfer Skin Tap Technique and ShotBlocker Technique, which are easy to apply and proven effective in reducing pain in infancy vaccination applications, are limited.

Therefore, this study aims to examine the effectiveness of the Helfer Skin Tap Technique and the ShotBlocker Technique in reducing pain in babies receiving intramuscular vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Born between 38 and 42 weeks of gestation,
* Between 2 and 4 months old,
* Applying to the family health center for KPA (Conjugated Pneumococcal Vaccine) application,
* No congenital anomalies, birth asphyxia or any chronic disease

Exclusion Criteria:

* Born prematurely or postmaturely
* Not between 2 and 4 months old
* Those who come to the family health center for the administration of other vaccines other than the KPA (Conjugated Pneumococcal Vaccine) application administered via IM route.
* Those with congenital anomalies, birth asphyxia or any chronic disease

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale = NIPS | Immediately after vaccination, the baby's pain will be evaluated with the Newborn Infant Pain Scale (NIPS).
  The Newborn-Infant Pain Scale, developed by Lawrence et al. (1993) to evaluate the physiological and behavioral responses of newborns to pain, was adapted into Turkish by Akdovan (1999). Scale; It consists of five behavioral and one physiological parts, including facial expression, crying, breathing pattern, arm and leg movements, and sleep-wake state. The crying part of the scale is given 0-1 and 2 points, and the other parts are given 0-1 point. The total score can range from 0 to 7, and a score higher than 3 indicates greater pain intensity.

IPD SHARING:
Plan to Share IPD: No